CLINICAL TRIAL: NCT04031417
Title: Modelling Endothelial Function With Hypoxia and Low Humidity (Simulated Flight Environment) in Healthy Volunteers and Patients With Type 2 Diabetes
Brief Title: Effect of a Simulated Flight in Patients With Type 2 Diabetes and Healthy Volunteers
Acronym: FlyBar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R1276
Record Dates: First submitted 2019-07-11; First posted 2019-07-24 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — SLH1 protein, Arabidopsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Other): Spend 2 hours in an environmental chamber at sea level conditions (temperature : 23c, oxygen concentration 21 %, humidity 45%) Spend 2 hours in a simulated flight (temperature 23c, oxygen concentration 15%, humidity 15%)
  Interventions: Other: Hypoxia; Other: Low Humidity
- soy isoflavones (Other): Spend 2 hours in an environmental chamber at sea level conditions (temperature : 23c, oxygen concentration 21 %, humidity 45%) Spend 2 hours in a simulated flight (temperature 23c, oxygen concentration 15%, humidity 15%)
  Interventions: Other: Hypoxia; Other: Low Humidity
- soy isoflavones & cocoa polyphenols (Other): Spend 2 hours in an environmental chamber at sea level conditions (temperature : 23c, oxygen concentration 21 %, humidity 45%) Spend 2 hours in a simulated flight (temperature 23c, oxygen concentration 15%, humidity 15%)
  Interventions: Other: Hypoxia; Other: Low Humidity

INTERVENTIONS:
Other: Hypoxia
Other: Low Humidity

SUMMARY:
Diabetes is an increasingly common condition which affects millions of people in the United Kingdom. Patients with type 2 diabetes are at increased risk to develop severe heart disease and vascular complications and these can result in death. A cornerstone of the treatment is lifestyle and diet.

The number of travellers is increasing quickly and there are more people than ever travelling by airplane. During a commercial flight the pressure of the air is lower than the pressure on the surface and that results in lower concentration of oxygen in the air we are breathing while flying. Also the humidity is very low inside an aircraft.

The aims of this study are to show if we can use a simulated flight as a method to look at how the endothelial cells react and to see if this is different between patients with type 2 diabetes mellitus and healthy volunteers.

A sub-study is also incorporated to look at different dietary interventions in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

Diabetes group:

* Diagnosis of type 2 diabetes
* Patients on stable medication (for their diabetes metformin being the only treatment if any), for 3 months prior to entry into the study
* Age between 45-75 years at the start of the study; women need to be postmenopausal and not undergoing hormone replacement therapy (HRT)

Healthy volunteers group:

* No current disease or medication which would have effect on the safety of the subjects or interfere with the study results
* Age between 45-75 years at the start of the study; women need to be postmenopausal and not undergoing HRT

Exclusion Criteria:

* For both groups:

  * Patients with concurrent illness or any medication in the last 3 months that would interfere with the study based on the investigator's judgement
  * Acute coronary syndrome in the last 3 months or any major clinical event in the previous 3 months that would effect the study based on the investigator's judgement
  * Patients not wishing to allow disclosure to their general practitioner (GP)s.
  * HbA1c >9%
  * Smokers
  * Pre-menopausal women or post-menopausal women on HRT
  * Claustrophobia, panic attacks in the anamnesis
  * Subjects must not have been subjected to a commercial flight within 4 weeks of the study

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Hypoxia and low humidity on the endothelial function in healthy volunteers and patients with type 2 diabetes using Wilcoxon signed rank test | Change from Baseline to 2 hours
  To determine the effect of hypoxia and low humidity on the endothelial function in healthy volunteers and patients with type 2 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Sathyapalan Thozhukat, MBBS MD, Principal Investigator — University of Hull, UK

REFERENCES:
- [Result] Konya J, Spurgeon BEJ, Al Qaissi A, Sathyapalan T, Ajjan R, Madden L, Naseem KM, Garrett AT, Kilpatrick E, Atkin SL. The Effect of a Simulated Commercial Flight Environment with Hypoxia and Low Humidity on Clotting, Platelet, and Endothelial Function in Participants with Type 2 Diabetes - A Cross-over Study. Front Endocrinol (Lausanne). 2018 Feb 13;9:26. doi: 10.3389/fendo.2018.00026. eCollection 2018. PMID 29487564
- See also: Publication Link — https://www.frontiersin.org/articles/10.3389/fendo.2018.00026/full